CLINICAL TRIAL: NCT00005805
Title: Does Hypericum Reduce Fatigue in Cancer Patients on Chemotherapy? A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: St. John's Wort in Relieving Fatigue in Patients Undergoing Chemotherapy or Hormone Therapy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: 99-102; MSKCC-99102; NCI-G00-1772
Record Dates: First submitted 2000-06-02; First posted 2004-07-26 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Myeloproliferative Disorders; Fatigue; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; childhood Burkitt lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; stage 0 chronic lymphocytic leukemia; Waldenström macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I small lymphocytic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage I adult non-Hodgkin lymphoma; stage II adult non-Hodgkin lymphoma; stage II small lymphocytic lymphoma; stage II grade 1 follicular lymphoma; stage II grade 2 follicular lymphoma; stage II grade 3 follicular lymphoma; stage II adult diffuse small cleaved cell lymphoma; stage II adult diffuse mixed cell lymphoma; stage II adult diffuse large cell lymphoma; stage II adult immunoblastic large cell lymphoma; stage II adult lymphoblastic lymphoma; stage II adult Burkitt lymphoma; stage III small lymphocytic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV small lymphocytic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; primary central nervous system non-Hodgkin lymphoma; fatigue; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; primary systemic amyloidosis; intraocular lymphoma; stage I mantle cell lymphoma; contiguous stage II adult non-Hodgkin lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult non-Hodgkin lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage II mantle cell lymphoma; multiple myeloma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; stage I marginal zone lymphoma; stage II marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Fatigue; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — Hypericum extract LI 160

INTERVENTIONS:
Dietary Supplement: St. John's wort

SUMMARY:
RATIONALE: Giving St. John's wort may be effective in relieving fatigue in patients with cancer who are undergoing chemotherapy or hormone therapy.

PURPOSE: Randomized phase III trial to determine the effectiveness of St. John's wort in relieving fatigue in patients who are undergoing chemotherapy or hormone therapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of Hypericum perforatum (St. John's Wort) in relieving fatigue in patients undergoing chemotherapy or hormonal therapy for malignant disease. II. Determine the relationship between fatigue, depression, and anxiety in these patients. III. Determine the correlation between quality of sleep and level of fatigue in these patients.

OUTLINE: This is a randomized, placebo controlled study. Patients are randomized to one of two treatment arms. Arm I: Patients receive oral Hypericum perforatum (St. John's Wort) 3 times a day. Arm II: Patients receive an oral placebo 3 times a day. Treatment continues for 6 weeks in the absence of worsening symptoms or unacceptable toxicity. Patients complete the Profile of Mood States (POMS) and the Brief Fatigue Inventory at the beginning and end of the study.

PROJECTED ACCRUAL: A total of 220 patients (110 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients with malignant disease receiving chemotherapy regimen for at least 6 weeks but less than 6 months, and continuing concurrent chemotherapy for at least 3-4 weeks OR Patients with malignant disease receiving hormonal therapy for at least 3 months prior to study, and continuing during entire study Profile of Mood States (POMS) Fatigue Subscale score of 14 or higher POMS Depression Subscale score of 13 or less

PATIENT CHARACTERISTICS: Age: Over 17 Performance status: Karnofsky 70-100% Life expectancy: At least 3 months Hematopoietic: Hemoglobin at least 10 g/dL No decline in hemoglobin of 2 g/dL or more for one month prior to study Hematocrit at least 30% Hepatic: SGOT no greater than 3 times upper limit of normal Bilirubin less than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No unstable cardiac disease Pulmonary: No debilitating pulmonary disease Other: No uncontrolled pain No uncontrolled serious infection No significant comorbidity that would preclude study participation Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: See Disease Characteristics Radiotherapy: Not specified Surgery: Not specified Other: At least 1 month since prior Hypericum perforatum (St. John's Wort) No other concurrent St. John's Wort No concurrent monamine oxidase inhibitors (e.g., furazolidone, isocarboxazid, meclobremide, phenelzine, procarbazine, selegiline, and tranylcypromine) No concurrent sympathomimetic amines (e.g., amphetamine, phenylpropanolamine, and pseudoephedrine) or other stimulants such as methylphenidate No concurrent serotonin reuptake inhibitors (e.g., fluoxetine, paroxetine, sertraline, venlafaxine, nefazodone, mirtazepine, buspirone, and trazodone) or tricyclic antidepressants (e.g., amitriptyline, clomipramine, desipramine, doxepin, imipramine, nortriptyline, and protriptyline) No concurrent serotonergic agents (e.g., lithium, meperidine, and dextromethorphan) No concurrent active treatment for anemia (e.g., transfusions or epoetin alpha)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Straus, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619